CLINICAL TRIAL: NCT04941378
Title: A Pilot, Single Dose, Open-Label Study of OTL38 Injection (OTL38) for Intra-Operative Imaging of Folate Receptor Positive Ovarian Cancer
Brief Title: OTL38 Injection (OTL38) for Intra-Operative Imaging of Folate Receptor Positive Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to sponsor request
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 11818
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- OTL 38 (Experimental): The study drug in question is an Investigational New Drug (IND), folate analog ligand conjugated with an indole cyanine green-like dye called OTL38. There will be a single dose of 0.025 mg/kg for intravenous injection over approximately 60 minutes, completed at least 1 hour prior to intraoperative imaging
  Interventions: Drug: OTL38; Device: intraoperative imaging camera system

INTERVENTIONS:
Drug: OTL38 — One time infusion of OTL38
Device: intraoperative imaging camera system — intraoperative imaging camera system

SUMMARY:
The primary objective of the study is to compare the performance of different camera imaging systems in assessing the positive predictive values and sensitivity of OTL38 to detect folate positive ovarian cancer cancers using the gold standard of pathologic review.

DETAILED DESCRIPTION:
Patients will be seen in the Ovarian Cancer Clinic. Patients that have or are suspected to have ovarian cancer, and are candidates for debulking surgery based on the clinician evaluation, may be considered candidates for this study. As over 90% of ovarian epithelial cancers express folate receptor, we would expect a high percentage of these patients scheduled for surgery, to have eligible cancer types for entry into the study. These patients will be prospectively consented to participate in this trial. There will be no randomization or control group and only patients previously scheduled to undergo surgery will be eligible to participate. We anticipate a 2-year period will be necessary to reach our accrual goal of up to 10 patients.

After obtaining informed consent, patients will receive a one-time dose of 0.025 mg/kg of OTL38, infused over approximately 60 minutes and completed at least 1 hour prior to intraoperative imaging. As a prophylactic measure, we recommend 25mg of IV Benadryl to the patient prior to the infusion of OTL38 to decrease the possibility of a hypersensitivity reaction.

The duration of surgical procedures to resect ovarian cancers varies substantially, anywhere from 3- 8 hours or more. During the phase 2 study, the median time spent imaging the patients with a single camera was 14 minutes. Utilizing two cameras to complete imaging would not overly increase the duration of time patients spend under anesthesia. However, there is a chance that being under anesthesia for the additional 25-35 minutes could put the patient at an increased risk of having of a common side effect associated with anesthesia. These common side effects include, but are not limited to: nausea and vomiting after surgery, sore throat and hoarseness, shivering/chills, confusion, and muscle aches

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years of age
* Have a primary diagnosis, or at high clinical suspicion, of primary ovarian cancer (of epithelial type), planned for primary surgical cytoreduction, interval debulking, or have recurrent ovarian cancer
* Good operative candidate as determined by clinical presentation and laboratory assessments
* Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

* Pregnant women as determined by urinary or serum beta hCG.
* Patients with a history of allergy to any of the components of OTL38, including folic acid
* Known FR-negative ovarian cancer
* Patients with a known allergy to Benadryl
* Previous exposure to OTL38
* Vulnerable populations: the homeless, prisoners or not capable of participating in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-28 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Compare the performance of different camera imaging systems in assessing the positive predictive values | Up to 4 weeks post surgery (completion of post-operative follow-up visit)
  The primary objective of the study is to compare the performance of different camera imaging systems in assessing the sensitivity and positive predictive value of OTL38 to detect folate positive ovarian cancers using the gold standard of pathologic review.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States